CLINICAL TRIAL: NCT02936609
Title: Assessing Community Cancer Care After Insurance ExpanSionS
Acronym: ACCESS
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: OCHIN, Inc. (Other); Health Choice Network (Other); Fenway Community Health (Other); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Devoe, MD, Principal Investigator, Oregon Health and Science University
Other Study IDs: 1R01CA204267 (NIH)
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Cancer
Keywords: healthcare access; healthcare utilization; preventive services; cancer survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Medicaid Expansion States: Patients receiving care in community health centers in states that expanded Medicaid (intervention group)
  Interventions: Other: Medicaid Expansion
- Medicaid Non-Expansion States: Patients receiving care in community health centers in states that did not expand Medicaid (control group)
  Interventions: Other: Medicaid Expansion

INTERVENTIONS:
Other: Medicaid Expansion — There will be no direct intervention, but rather an observation of change based on whether a state expanded Medicaid or not

SUMMARY:
This innovative and timely study will measure the impact of Affordable Care Act (ACA) Medicaid expansions on cancer screenings and preventive services. To assess this natural policy experiment, the investigators will use electronic health record data from the Accelerating Data Value Across a National Community Health Center Network (ADVANCE) clinical data research network (CDRN) of the National Patient-Centered Clinical Research Network (PCORnet).

DETAILED DESCRIPTION:
Cancer morbidity and mortality is greatly reduced through screening and prevention, but uninsured patients are much less likely than insured patients to receive these evidence-based services as recommended. In addition, uninsured cancer survivors receive fewer primary and preventive care services than those with health insurance. Thus, it is hypothesized that Affordable Care Act (ACA) Medicaid expansions could substantially improve access to essential cancer preventive and screening services for previously uninsured patients, and facilitate better care for cancer survivors who gain health insurance. In 2012, the United States (US) Supreme Court ruled that states were not legally required to implement ACA Medicaid expansions, creating a unique natural experiment to test this hypothesis. By April 1, 2015, 30 states and the District of Columbia had implemented expansions, and 20 states had not. This led to increased Medicaid enrollment by 26% in expansion states, compared to 8% in non-expansion states. Previous single-state Medicaid expansions led to increased utilization of healthcare services and improved health outcomes post-expansion. For example, in Oregon, cervical cancer screening rates were 18-19% higher among women who gained Medicaid in 2008, compared to those who remained uninsured. However, no previous assessments of state-specific expansions had concurrent control (non-expansion) states for comparison. Further, little is known about how Medicaid expansion impacts the delivery of recommended primary and preventive care services to cancer survivors, termed 'survivor care.'

The investigators propose to use the ACA Medicaid expansion natural experiment to study the effect of state-level Medicaid expansion on rates of cancer screening and preventive services ('cancer prevention') and survivor care. Many patients likely to gain coverage through ACA Medicaid expansions receive primary care in community health centers (CHCs), our nation's healthcare 'safety net;' thus, the proposed analyses will use electronic health record (EHR) data from the ADVANCE clinical data research network (CDRN) of CHCs (ADVANCE is one of 11 CDRNs in the national PCORnet data network). The ADVANCE CDRN has patient-level data from 476 CHCs in 13 Medicaid expansion states (n=576,711 patients) and 242 CHCs in 8 non-expansion states (n=361,421 patients). This nationally unique data resource will allow us to measure outcomes in expansion versus non-expansion states, illuminating the impact of increased Medicaid opportunities on rates of cancer prevention and survivor care within the safety net. The investigators will also assess whether disparities in delivery of this care are reduced. Our specific aims for this study, titled "Assessing Community Cancer care after insurance ExpanSionS (ACCESS)," are to:

Aim 1. Compare pre-post receipt of cancer prevention and screening among vulnerable CHC patients in Medicaid expansion versus non-expansion states.

Hypothesis 1a: Cancer prevention and screening will significantly increase among CHC patients in expansion states, compared to those in non-expansion states.

Hypothesis 1b: Racial/ethnic disparities in cancer prevention and screening will be significantly reduced in expansion states versus no change in non-expansion states.

Aim 2. Compare pre-post insurance status, visits, and receipt of routine, recommended primary and preventive care among cancer survivors seen in CHCs in expansion versus non-expansion states.

Hypothesis 2a: A higher percentage of uninsured cancer survivors will have gained insurance coverage in expansion states, compared to those in non-expansion states.

Hypothesis 2b: Cancer survivors who are CHC patients in expansion states will have a significant increase in visits, visits paid by Medicaid, and survivor care relative to no change among patients in non-expansion states.

ELIGIBILITY:
Inclusion Criteria:

* Patients in intervention and control states aged 19-64

Exclusion Criteria:

* Patients at intervention and control clinics outside of the age range 19-64

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study eligible patients within electronic health record data from the ADVANCE CDRN of PCORnet
Sampling Method: Non-Probability Sample
Enrollment: 1939783 (Actual)
Dates: Start 2016-04; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Change in number of preventive services received | Less than or equal to 24 months prior to Medicaid expansion vs greater than or equal to 24 months post
  Preventive services and screenings for cervical, colorectal, and breast cancers, HPV vaccinations, smoking screening ad interventions, and obesity screening and interventions.

SECONDARY OUTCOMES:
Change in type of preventive services received | Less than or equal to 24 months prior to Medicaid expansion vs greater than or equal to 24 months post
  Preventive services and screenings for cervical, colorectal, and breast cancers, HPV vaccinations, smoking screening ad interventions, and obesity screening and interventions
Change of health insurance status | Less than or equal to 24 months prior to Medicaid expansion vs greater than or equal to 24 months post
  Health insurance status derived from EHR data and is primarily based on information collected at each visit
Change in number of primary care visits | Less than or equal to 24 months prior to Medicaid expansion vs greater than or equal to 24 months post
  Number of primary care visits.
Change in type of primary care visits | Less than or equal to 24 months prior to Medicaid expansion vs greater than or equal to 24 months post
  Types of primary care visits.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bailey SR, Marino M, Ezekiel-Herrera D, Schmidt T, Angier H, Hoopes MJ, DeVoe JE, Heintzman J, Huguet N. Tobacco Cessation in Affordable Care Act Medicaid Expansion States Versus Non-expansion States. Nicotine Tob Res. 2020 May 26;22(6):1016-1022. doi: 10.1093/ntr/ntz087. PMID 31123754
- [Result] Hoopes M, Schmidt T, Huguet N, Winters-Stone K, Angier H, Marino M, Shannon J, DeVoe J. Identifying and characterizing cancer survivors in the US primary care safety net. Cancer. 2019 Oct 1;125(19):3448-3456. doi: 10.1002/cncr.32295. Epub 2019 Jun 7. PMID 31174231
- [Result] Hoopes M, Voss R, Angier H, Marino M, Schmidt T, DeVoe JE, Soule J, Huguet N. Assessing Cancer History Accuracy in Primary Care Electronic Health Records Through Cancer Registry Linkage. J Natl Cancer Inst. 2021 Jul 1;113(7):924-932. doi: 10.1093/jnci/djaa210. PMID 33377908
- [Result] Huguet N, Angier H, Rdesinski R, Hoopes M, Marino M, Holderness H, DeVoe JE. Cervical and colorectal cancer screening prevalence before and after Affordable Care Act Medicaid expansion. Prev Med. 2019 Jul;124:91-97. doi: 10.1016/j.ypmed.2019.05.003. Epub 2019 May 8. PMID 31077723
- [Result] Angier HE, Marino M, Springer RJ, Schmidt TD, Huguet N, DeVoe JE. The Affordable Care Act improved health insurance coverage and cardiovascular-related screening rates for cancer survivors seen in community health centers. Cancer. 2020 Jul 15;126(14):3303-3311. doi: 10.1002/cncr.32900. Epub 2020 Apr 15. PMID 32294251
- [Derived] Angier H, Huguet N, Marino M, Mori M, Winters-Stone K, Shannon J, Raynor L, Holderness H, DeVoe JE. Assessing Community Cancer care after insurance ExpanSionS (ACCESS) study protocol. Contemp Clin Trials Commun. 2017 Sep;7:136-140. doi: 10.1016/j.conctc.2017.06.011. Epub 2017 Jun 24. PMID 29473059